CLINICAL TRIAL: NCT06273865
Title: Version Testing of EnzySystem Version A for Hemophilia A
Status: Suspended | Type: Observational
Why Stopped: Performing interim analysis before continuing with next center
Sponsor: Radboud University Medical Center (Other)
Collaborators: Enzyre B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMSTOL77
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-08

CONDITIONS: Hemophilia A
Keywords: Diagnostic; Point of care; Thrombin generation; Factor VIII
MeSH Terms: conditions — Hemophilia A; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples for reference assays and additional coagulation tests will be centrifuged at 4°C (3000g, 10 min) to obtain plasma. Red blood cells and platelets are discarded.
  Plasma of the venipuncture will be aliquoted in portions of 250 µL, snap frozen in liquid nitrogen or frozen using dry ice, and stored at -80°C. All steps until freezing of the plasma should take place within two hours after venipuncture. Samples are stored until the data of this study has been published, but not longer than 5 years. After consent of the participant samples can be stored for 15 years maximally to use for analyses of other studies from Enzyre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy volunteers
  Interventions: Diagnostic Test: Several assays
- Hemophilia A patient
  Interventions: Diagnostic Test: Several assays

INTERVENTIONS:
Diagnostic Test: Several assays — Standard blood draw by venipuncture is performed in all study participants to collect blood samples in four 2.7 mL citrated blood tubes. Tube one is a dummy tube and is discarded. Tube two is used for the FVIII activity and thrombin generation assay on the EnzySystem. Tube three is used to perform conventional FVIII activity and thrombin generation assays. Tube four is used for duplicate measurements of the conventional assays and measurement of prothrombin F1+2 antigen levels, ADAMTS13 activity, FVIII antigen, VWF (von Willebrand Factor) antigen and von Willebrand ristocetin cofactor activity levels.

SUMMARY:
Background of the study:

To measure blood clotting, blood is taken from a vein. This blood is processed in the laboratory and then tested. A new device has been developed that requires only a very small volume of blood (5-10 drops of blood) to perform the laboratory tests. The long-term goal is that this device can be used by a doctor or at home to quickly measure blood clotting. In this research we want to compare this new system with the standard methods - measurement in the laboratory - and evaluate whether the correct value is determined.

Objective of the study:

The primary objective of this study is to demonstrate that the EnzySystem HemA version A can record thrombin generation TG and quantify FVIII activity levels within a time frame of 60 min in fresh whole blood samples of healthy volunteers and patients with hemophilia A in the Enzyre laboratory (for healthy volunteers) and the Radboudumc (for patients with hemophilia A).

Study design:

This is a cross-sectional observational study. All participants are asked to fill a questionnaire prior to blood collection. The blood of healthy volunteers will be collected in an office of Enzyre BV, the blood of patients will be collected in the Radboudumc. Blood collection, by venepuncture, will be conducted by a Radboudumc research nurse or physician of the research team in both locations. In total, four blood tubes with citrate as anticoagulant will be drawn (a total of around 11 mL).

Study population:

The study population consists of 20 healthy volunteers: evenly distributed between male and female; ages spread over the range from 20 to 70 years old; recruited by Enzyre via advertisement. 20 Patients: 5 severe hemophilia A; 5 moderate hemophilia A; 10 mild hemophilia A; recruited from the Hemophilia Treatment Center (HTC) Nijmegen-Eindhoven-Maastricht (NEM) (location Radboudumc).

Primary study parameters/outcome of the study:

Demonstrate that the EnzySystem HemA version A can record TG and quantitative FVIII activity levels within a time frame of 60 min in fresh blood samples of healthy volunteers and patients with hemophilia A.

Secondary study parameters/outcome of the study (if applicable):

Secondary study parameters are composed whether the measured values comply with the desired assay specificity and accuracy.

Outcomes are analysed for equivalence compared to one-stage FVIII assay, FVIII chromogenic assay, thrombin generation via the Nijmegen Hemostasis Assay, and possibly via the Technoclone assay.

Is it possible to measure FVIII activity with the EnzySystem HemA version A in fresh blood samples of healthy volunteers and patients with hemophilia A, compared to the gold standard with;

* Precision in the normal range (60-140%): min. 30%
* Precision in the low range (3-10%): min. 50%
* Limit of Detection range min. 100 % FVIII activity
* Limit of Detection low range min. 3 % FVIII activity Is it possible to measure TG with the EnzySystem HemA version A in fresh blood samples of healthy volunteers and patients with hemophilia A, compared to the gold standard with;
* Precision in the normal range (60-140%) of control samples: min. 30%
* Precision in patient with hemophilia A: min. 50%
* Limit of Detection, high range > 400 nM thrombin activity
* Limit of Detection measured with Plasma, low range < 50 nM thrombin

Other study parameters All samples will also be tested for other hemostasis specific parameters as these parameters may affect a proper measurement of both FVIII activity and Thrombin Generation. The following parameters will be measured in plasma obtained from the whole blood vacutainers. Moreover, left over samples (plasma) will eventually be used to develop other coagulation related parameters.

* von Willebrand Factor antigen levels
* von Willebrand Factor ristocetin activity levels
* Prothrombin Fragment 1+2 levels
* ADAMTS13 activity
* FVIII antigen levels
* blood group

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Age between 20 to 70 years old (equally distributed over the age range)
* 7 volunteers 20-40 years old
* 7 volunteers 40-60 years old
* 6 volunteers 60+ years old

Hemophilia A patients:

* Diagnosed with mild (FVIII activity levels 5-40%), moderate (FVIII activity levels 1-5%) or severe hemophilia A (FVIII activity levels <1%)
* Medication

  1. On demand treatment
  2. Washout of medication of at least 24 hours after treatment with short half life (SHL) replacement therapy
  3. Washout of medication of at least 72 hours after treatment with extended half life (EHL) replacement therapy
* Age 20-70 years old

Exclusion Criteria:

A healthy volunteer who meets any of the following criteria will be excluded from participation in this study:

* use of anticoagulants or platelet antagonists (aspirin or any TAR);
* known allergy to stainless steel;
* trauma or surgery within the last two weeks;
* pregnancy;
* use of:

  * NSAIDs;
  * antimicrobial medication;
  * thyroid inhibitors; or SSRI's. A hemophilia A patient who meets any of the following criteria will be excluded from participation in this study:
* use of anticoagulants or platelet antagonists (aspirin or any TAR);
* known allergy to stainless steel;
* trauma or surgery within the last two weeks;
* a bleeding episode within the last two weeks;
* clinical indication of liver cirrhosis (echographic indication, enlarged spleen, decreased platelet count);
* pregnancy;
* FVIII inhibitors;
* Signs of inflammation or infection
* use of:

  * NSAIDs;
  * antimicrobial medication;
  * thyroid inhibitors or SSRI's;
  * Emicizumab.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy volunteers who respond to an advertisement at the Noviotech campus in Nijmegen
  Hemophilia A patients are recruited from the Hemophilia Treatment Center (HTC) Nijmegen-Eindhoven-Maastricht (NEM) (location Radboudumc).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Time between venipuncture and EnzySystem assay results | All measurements with the EnzySystem will be performed <2 hours of drawing blood
  Time is measured between venipuncture, start of the EnzySystem FVIII activity and thrombin generation assay, and assay results

SECONDARY OUTCOMES:
Validity of EnzySystem FVIII activity results | All steps until freezing of the plasma should take place within two hours after venipuncture
  Comparison of the FVIII activity results obtained with the EnzySystem and with conventional (one-stage and chromogenic) assays
Validity of EnzySystem thrombin generation results | All steps until freezing of the plasma should take place within two hours after venipuncture
  Comparison of the thrombin generation results obtained with the EnzySystem and with conventional assays

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Schols, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Enzyre BV, Nijmegen, Gelderland
  - Radboud university medical center, Nijmegen

IPD SHARING:
Plan to Share IPD: No